CLINICAL TRIAL: NCT04146194
Title: OTTAPE : Observatory on the Use of New Therapies (LED Photobiomodulation, Radiofrequency, Laser and Injectable Hyaluronic Acid) in the Treatment of Women's Pelvic-perineal Pathologies After Failure, Partial or Total, of First-line Medical Treatment
Acronym: OTTAPE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018/PM-01; 2019-A00665-52 (Other: ANSM)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-02

CONDITIONS: Pelvic-perineal Pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None. This is a non-interventional observational study. — None. This is a non-interventional observational study.

SUMMARY:
Women's pelvic-perineal pathologies are a very frequent reason for consultation in gynaecology. The symptoms reported are diverse and range from the most frequent (genital prolapse, urinary or anal incontinence, dysuria, chronic pain) to new complaints (dyspareunia, vaginal laxity, perineum scarring, vulvo-vaginal atrophy).

Currently, first-line medical treatments are no longer sufficient to improve patients. New therapies have emerged, namely LED photobiomodulation, radio frequency, Erbium or fractionated CO2 laser and injectable hyaluronic acid.

These new treatments have been used in common practice for several years, but no studies have standardized practices. There are no recommendations regarding these new therapies to give specific indications for their use.

The aim is to standardise the indications for these new technologies.

* LED photobiomodulation: management of scar perineas with pain, scarring disorders or trophic disorders.
* The Erbium laser or fractionated CO2: treatment of vulvo-vaginal atrophy.
* radiofrequency: management of chronic pelvic-perineal and postpartum pain.
* injectable hyaluronic acid: treatment of vestibulodynia and trophic disorders. Non-validated indications are proposed for these therapies (urinary incontinence, vaginal laxity and prolapse)

DETAILED DESCRIPTION:
Initially, this involves the follow-up of patients treated in the Gynaecology-Obstetrics department of the University Hospital of Nîmes and the Karis medical centre of Perpignan for a pelvi-perineal pathology. Other centres will be gradually incremented. Patients will have received a letter of information and no objection to the prospective collection of her data as part of routine management without any other intervention. These patients should not have any contraindications to the use of these new therapies.

At inclusion, the patient receives a pelvic-perineal clinical examination and a functional assessment (vaginal sampling), pain (EVA). The FSFI questionnaire will be administered.

During this visit, the investigator will set up a treatment with a new therapy. This treatment will be chosen by the operator before recommendations are made. The operator must detail the type of device and the protocol chosen.

The patient will be reviewed 4 weeks after the end of her treatment: she will benefit from an evaluation identical in all respects to the inclusion visit with the administration of the PGI-I questionnaire.

All information concerning the discontinuation, continuation or change of treatment will be documented in this follow-up phase.

In case of failure, second line treatment may be offered. Possible adverse reactions will be collected at all times.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pelvic-perineal pathology
* Patients who are not opposed to prospective data collection.

Exclusion Criteria:

* Patients with contraindications to these new therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initially, this involves the follow-up of patients treated in the Gynaecology-Obstetrics department of the University Hospital of Nîmes and the Karis medical centre of Perpignan for a pelvi-perineal pathology. Other centres will be gradually incremented. Patients will have received a letter of information and no objection to the prospective collection of her data as part of routine management without any other intervention. These patients should not have any contraindications to the use of these new therapies.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Characteristics of patients who are candidates for these new therapies | 12 month
  Set up an observatory to carry out an inventory of the use of these new technologies and provide answers to basic questions: who uses them, for which patients, in which indications and for which therapeutic gain? Collect the practices of professionals and make it possible to evaluate the effectiveness of the therapeutic choice by the physician and the patient.
First-line treatment tried | 12 month
  Set up an observatory to carry out an inventory of the use of these new technologies and provide answers to basic questions: who uses them, for which patients, in which indications and for which therapeutic gain? Collect the practices of professionals and make it possible to evaluate the effectiveness of the therapeutic choice by the physician and the patient.
Type of therapy used and for which type of pathology | 12 month
  Set up an observatory to carry out an inventory of the use of these new technologies and provide answers to basic questions: who uses them, for which patients, in which indications and for which therapeutic gain? Collect the practices of professionals and make it possible to evaluate the effectiveness of the therapeutic choice by the physician and the patient.
Number of sessions performed | 12 month
  Set up an observatory to carry out an inventory of the use of these new technologies and provide answers to basic questions: who uses them, for which patients, in which indications and for which therapeutic gain? Collect the practices of professionals and make it possible to evaluate the effectiveness of the therapeutic choice by the physician and the patient.
Possible use of a second therapy | 12 month
  Set up an observatory to carry out an inventory of the use of these new technologies and provide answers to basic questions: who uses them, for which patients, in which indications and for which therapeutic gain? Collect the practices of professionals and make it possible to evaluate the effectiveness of the therapeutic choice by the physician and the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forret A, Mares P, Delacroix C, Chevallier T, Potier H, Fatton B, Masia F, Ripart S, Letouzey V, de Tayrac R, Salerno J. [Photobiomodulation and vulvovaginal disorders after anticancer treatments]. Bull Cancer. 2023 Sep;110(9):883-892. doi: 10.1016/j.bulcan.2023.03.018. Epub 2023 May 12. French. PMID 37183056